



# TARGETING MICROENVIRONMENT AND CELLULAR IMMUNITY IN SARCOMAS WEEKLY TRABECTEDIN COMBINED WITH METRONOMIC CYCLOPHOSPHAMIDE IN PATIENTS WITH ADVANCED PRETREATED SOFTTISSUE SARCOMAS A PHASE I/II STUDY FROM THE FRENCH SARCOMA GROUP

# **Protocol TARMIC**

VERSION N°6.0 DU |11|12|2018|- N°: IB 2015-04

Intégrant la modification substantielle n°1 du 20/01/2016 Intégrant la modification substantielle n°2 du 28/10/2016 Intégrant la modification substantielle n°3 du 26/04/2017 Intégrant la modification substantielle n°4 du 19/10/2017 Intégrant la modification substantielle n°5 du 11/12/2018

# EudraCT n° 2015-002760-16

# **Coordinating Investigator**

Antoine ITALIANO, MD, PhD *Medical Oncologist* 

Department of Medical Oncology Institut Bergonié

229, cours de l'Argonne – 33076 BORDEAUX Cedex, France

Tél: 05.56.33.78.05 - Fax: 05.56.33.04.85 - E-mail: a.italiano@bordeaux.unicancer.fr

#### **Clinical Research Unit**

Simone MATHOULIN-PÉLISSIER, MD, PhD

Responsable UREC

Marina PULIDO, MsC

Biostatisticien, UREC

Sabrina SELLAN-ALBERT, MsC

Attachée de Recherche Clinique, UREC

Institut Bergonié, Bordeaux

Institut Bergonié, Bordeaux

Institut Bergonié, Bordeaux

# Pharmacist and Vigilance Unit

Emilie TOULZA, PharmD

Institut Bergonié, Bordeaux

**SPONSOR** 

**INSTITUT BERGONIE** 

# APPROVAL AND SIGNATURES OF PROTOCOL

**Protocol title**: Targeting Microenvironment and Cellular Immunity in Sarcomas Weekly trabectedin combined with Metronomic Cyclophosphamide in Patients with Advanced Pretreated Soft-tissue Sarcomas. A Phase I/II study from the French Sarcoma Group.

| | | Date de l'autorisation initiale | 19/10/2015 |
|---|---|---|---|
| | | Autorisation de la modification substantielle 1 | 10/03/2016 |
| | | Autorisation de la modification substantielle 2 | 29/12/2016 |
| Competent | Name : ANSM | Autorisation de la modification substantielle 3 | 13/10/2017 |
| authority | | Autorisation de la modification substantielle 4 | 02/05/2018 |
| | | Autorisation de la modification substantielle 5 | 06/02/2019 |
| | | Référence: | 151077A-12 |
| | | Date de l'avis favorable initial | 30/09/2015 |
| | | Autorisation de la modification substantielle 1 | 24/02/2016 |
| E4L* | Name: CPP du Sud-Ouest et d'Outre-Mer III | Autorisation de la modification substantielle 2 | 30/11/2016 |
| Ethic<br>Committee | | Autorisation de la modification substantielle 3 | 31/05/2017 |
| | | Autorisation de la modification substantielle 4 | 31/01/2018 |
| | | Autorisation de la modification substantielle 5 | 27/02/2019 |
| | | Référence : | 2015/94 |

| Name and responsability | Address | Date | Signature |
|---|---|---|---|
| Managing Director | Pr François-Xavier MAHON<br>Institut Bergonié – Bordeaux<br>Tél:05.56.33.33.33 / Fax: 05.56.33.33.30<br>Mail: f.mahon@bordeaux.unicancer.fr | 11/12/2018 | |
| Coordinating<br>Investigator | Pr Antoine ITALIANO Institut Bergonié – Bordeaux Tél 05.56.33.78.05 / Fax : 05.56.33.04.85 Mail : a.italiano@bordeaux.unicancer.fr | 11/12/2018 | A |
| Clinical Research<br>Manager | Pr Simone MATHOULIN-PÉLISSIER<br>Institut Bergonié – Bordeaux<br>Tél:05.56.33.33.98 / Fax: 05.56.33.04.66<br>Mail : s.mathoulin@bordeaux.unicancer.fr | 11/12/2018 | |
| Biostatistician | Marina PULIDO<br>Institut Bergonié – Bordeaux<br>Tél:05.24.07.19.29/Fax: 05.24.07.19.49<br>Mail : m.pulido@bordeaux.unicancer.fr | 11/12/2018 | # |
| Clinical Research<br>Assistant | Sabrina SELLAN-ALBERT<br>Institut Bergonié – Bordeaux<br>Tél:05.56.33.78.05/Fax:05.56.33.04.85<br>Mail : s.albert@bordeaux.unicancer.fr | 11/12/2018 | Selland |
| Pharmacist | Emilie TOULZA<br>Institut Bergonié – Bordeaux<br>Tél:05.47.30.60.53/Fax: 05.56.33.04.85<br>Mail: e.toulza@bordeaux.unicancer.fr | 11/12/2018 | |

I acknowledge having read the whole protocol, and I pledge to lead this protocol in accordance with the Good Clinical Practice (decision of 24 November 2006), the Public Health Law No. 2006-806 of August 09, 2004 and the implementing Decree  $n^{\circ}$  2006-477 of April 26, 2006 and as described in this document.

I assume my responsibilities as referent investigator including:

- Collection of informed consent, dated and signed by patients before any selection procedure in the protocol,
- Validation of case report forms, completed for each patient included in the study,
- Direct access to source documents for verification by the clinical research assistant (CRA) commissioned by the sponsor,
- Archiving of critical documents of the study for a 15 year-period.

| Name and address of the hospital | |
|----------------------------------------|------------|
| Name of the Coordinating Investigator: | |
| Date : | Signature: |

| Title of the study | Targeting Microenvironment and Cellular Immunity in Sarcomas Weekly trabectedin combined with Metronomic Cyclophosphamide in Patients with Advanced Pretreated Soft-tissue Sarcomas. A Phase I/II study from the French Sarcoma Group |
|---|---|
| Abbreviation of the trial | TARMIC |
| <b>Sponsor Identification</b> | Institut Bergonié, Regional Comprehensive Cancer Center |
| Coordinating | Professor Antoine ITALIANO |
| Number of investigational sites planned | Department of Medical Oncology Phase I: 1 centre - Institut Bergonié Phase II: 1 centre - Institut Bergonié |
| Number of patients | Phase I: 12 - 24 patients Phase II: 47 patients |
| Duration of the study | Planned enrollment period: 48 months Treatment duration: until progression Follow-up: 12 months Study period: 5 years |
| <b>Medical conditions</b> | Adult patients with unresectable locally advanced or metastatic soft-tissue sarcoma |
| Study design | Phase I: Monocentric Phase I trial based on a dose escalation study design (3+3 traditional design). Phase II: One-arm, monocentric Phase II trial based on two-stage optimal Simon's design. |
| Objectives | <ul> <li>Phase I: Primary objective: <ul> <li>To establish the recommended phase II dose (RP2D), the maximum tolerated dose (MTD) evaluated on the first cycle (D1 to D28), the safety profile, and the dose limiting toxicities (DLT) of trabectedin given in combination with CP.</li> </ul> </li> <li>Secondary objectives: <ul> <li>To evaluate preliminary signs of antitumor activity of trabectedin given in combination with CP in terms of objective response under treatment (as per RECIST v1.1 criteria), 6-month non-progression (as per RECIST v1.1 criteria), 1-year progression-free survival (PFS) (as per RECIST v1.1 criteria) and 1-year overall survival (OS).</li> <li>To describe the pharmacokinetics (PK) of trabectedin given in combination with CP.</li> <li>Biomarker study: To perform pharmacodynamic (PD)/mechanism of action (MOA) biomarkers analysis as well as predictive biomarkers analysis (levels of angiogenic and immunologic biomarkers in blood at baseline and different study time points).</li> <li>Ancillary study: To assess pharmacodynamics changes of Tissue Associated Macrophage (TAM) infiltration and additional tumor markers on fresh pre-treatment and on-treatment tumor biopsies.</li> </ul> </li> <li>Phase II: <ul> <li>Primary objective:</li> </ul> </li> <li>To evaluate the antitumor activity of trabectedin in association with CP in terms of non-progression at 6 months (complete or partial responses or stable disease more than 24 weeks, as per RECIST v1.1 criteria) after centralized radiological review, in patients with advanced STS who already failed anthracycline-containing chemotherapy (CT).</li> </ul> <li>Secondary objectives: <ul> <li>To evaluate the antitumor activity of trabectedin in association with CP in terms of objective response under treatment (as per RECIST v1.1 criteria), 1-year progression free survival (PS)</li></ul></li> |

| | Optional ancillary study: To assess pharmacodynamics changes of TAM infiltration and |
|---|---|
| | additional tumor markers on fresh pre-treatment and on-treatment tumor biopsies. |
| | 1 Deticate with a feeting account histolesis llarge found has control assistant (De Caindre |
| | 1. Patients with soft-tissue sarcoma histologically confirmed by central review (Pr. Coindre team), except in case of diagnosis was already confirmed by the RRePS Network, |
| | 2. Metastatic or unresectable locally advanced disease, |
| | 3. Age ≥ 18 years, |
| | 4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2, |
| | 5. Life expectancy > 3 months, |
| | 6. Measurable disease according to RECIST v1.1 (lesion in previously irradiated field can be |
| | considered as measurable if progressive at inclusion according to RECIST v1.1), |
| | 7. For patients included in phase II study, progressive disease according to RECIST v1.1 criteria |
| | diagnosed on the basis of two CT scan or MRI obtained at an interval less than 6 months in the |
| | period of 12 months prior to inclusion and confirmed by central review. PET-CT are also |
| | acceptable (two PET-CT or a CT scan compared with a PET-CT), under the following |
| | conditions: |
| | a. Target lesions must be evaluable on PET-CT according to RECIST v1.1. This will be |
| | determined by the central radiologist at the time of the review. If target lesions are not |
| | evaluable according to RECIST v1.1, patient will not be eligible. |
| | b. PET-CT is acceptable only for the central review. If not available, an additional CT scan |
| | (or MRI) must be performed within four weeks prior to Day 1 of cycle 1 (+1 week |
| | tolerance) to be used as baseline tumor assessment. Patient must be then followed using |
| | the same technique throughout the duration of the protocol, |
| | 8. Previous use of Anthracyclines, |
| | 9. Have provided tissue from an archival tissue sample, |
| | 10. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological |
| | treatment and/or radiotherapy, |
| Inclusion criteria | 11. Adequate hematological, renal, metabolic and hepatic function: |
| metasion eriteria | a. Hemoglobin ≥ 9 g/dl (patients may have received prior red blood cell [RBC] |
| | transfusion, if clinically indicated); absolute neutrophil count (ANC) $\geq 1.5 \times 10^9$ /l, |
| | leukocyte count $\geq 2.5 \times 10^9$ /l and platelet count $\geq 100 \times 10^9$ /l |
| | b. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) $\leq 2.5$ x upper limit |
| | of normality (ULN) ( $\leq 5$ in case of extensive liver involvement) and alkaline phosphatase |
| | $(AP) \le 2.5 \text{ x ULN}$ |
| | c. Total bilirubin ≤ ULN. d. Albumin ≥ 25 g/l |
| | e. Serum Creatinine $\leq 1.5$ x ULN or calculated creatinine clearance (CrCl) $\geq 30$ ml/min |
| | (according to Cockroft formula). |
| | f. Creatine Phosphokinase (CPK) $\leq 2.5 \text{ x ULN}$ |
| | 12. Women of childbearing potential must have a negative serum pregnancy test before study |
| | entry. Both women and men must agree to use a medically acceptable method of contraception |
| | throughout the treatment period and for six months after discontinuation of treatment. |
| | Acceptable methods of contraception include intrauterine device (IUD), oral contraceptive, |
| | subdermal implant and double barrier, |
| | 13. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for |
| | adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in |
| | situ transitional bladder cell carcinoma, |
| | 14. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment |
| | (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2) according to |
| | the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, |
| | version 4.0), |
| | 15. Patients with a social security in compliance with the French law, |
| | <ul><li>16. Voluntarily signed and dated written informed consent prior to any study specific procedure.</li><li>1. Previous treatment with Trabectedin,</li></ul> |
| | 2. Currently active bacterial or fungus infection (> grade 2 CTC [CTCAE]), HIV1, HIV2, |
| | hepatitis B or hepatitis C infections, |
| | 3. History of chronic alcohol use and/or cirrhosis, |
| Non Inclusion criteria | 4. The following unstable cardiac conditions are not allowed: |
| | - Congestive heart failure |
| | - Angina pectoris |
| | - Myocardial infarction within 1 year before registration |
| | , |

| | T.T., | 4 | 4.641.1. | | - > 150/100I | [ | 1 |
|---|---|---|---|---|---|---|---|
| | medical thera | ed arterial hypertensio | on defined as bio | oa pressur | e ≥ 150/100 mmF | ig despite opt | ımaı |
| | | ъру<br>s clinically significan | t | | | | |
| | | able to receive cortic | | | | | |
| | | ntral nervous system i | | S), | | | |
| | | women of childbear | | | ot using an effe | ective metho | d of |
| | | as previously describ | | | | | |
| | 8. Participation | on to a study involvin | g a medical or th | nerapeutic | intervention in the | e last 30 days | , |
| | | nrolment in the presen | | | | | |
| | | nable to follow and co | omply with the s | tudy proce | edures because of | any geograph | nical, |
| | | chological reasons, | | | 6: 6 1 : | | |
| | | ypersensitivity to any accination (in the last | | | | n component | s. |
| | | rinary tract obstructio | | iliciusioii) | ioi yenow ievei. | | |
| | 14. Cardiac d | | ·11. | | <b>A</b> | | |
| | | eft Ventricular Ejection | on Fraction) < 4 | 0% at base | eline: | | |
| | - or clinically symptomatic cardiac dysfunction (any % of LVEF at baseline) | | | | | | |
| | Cyclophosphamide will be administered bi-daily (50 mg x 2), and given on a week on/week off | | | | | | |
| Route of | schedule. Trabectedin will be administered by intravenous 3-hour infusion weekly for three consecutive | | | | | | |
| administration | | | | | | | |
| | | 1, 8 and 15) every 4 v | veeks. | | | | |
| | Phase I: Dose escalation part | | | | | | |
| | | <u> </u> | Regimen Descr | ription | | 6.1 | |
| | Agent | Premedication | Dose | Route | Schedule | Cycle<br>Length | |
| | | domperidone, | | | | Length | - |
| | CP | metoclopramide, | 50mg x 2 | per os | 1 week on /1 | 1 | |
| | | setrons allowed | | • | week off | | |
| | | 4 | Doses as | | Days 1, 8 and | 4 weeks | |
| | Trabected | 20 mg | appropriate | IV | 15 every 4 | + weeks | |
| | in | dexamethasone | for assigned | 1 | weeks | | |
| Treatment schedule | | 1 64 | dose level | | | | 1 |
| | A treatment cycle consists of 4 weeks. Treatment may continue until disease progression or | | | | | | |
| | study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.) | | | | | | |
| | Patients will be allocated to 4 doses of Trabectedin following a 3 + 3 design: | | | | | | |
| | Level -1 1 2 3 4 | | | | | | |
| | Trab | pectedin (mg/m²) - (3h | 1) 0.25 | 0.3 | 0.4 0.5 | 0.6 | |
| | Di Ti | | 1 1 . DD2D | C . 1 . | 1: 1 6: 1: .1 | | |
| | | patients will be treate<br>n association with me | | | | | |
| | phase I trial. | ii association with me | enonomic cyclop | люѕрпанн | de with the same | schedule as il | ii tiie |
| | Annennen votoctor | -limiting toxicities wi | ll be assessed fo | r 4 weeks. | | | |
| Safety and efficacy | 70000 | ll be assessed on Day | | | | | |
| evaluations | | be assessed every 2 c | | | | | |
| | Phase I trial: | | | | | | |
| | | ctive of the phase I tr | | | | | |
| | maximum tolerated doses (MTD) evaluated on the first cycle (D1 to D28), the safety profile, | | | | | | |
| | and the dose limiting toxicities (DLT) of trabectedin given in association with metronomic | | | | | | |
| | | | (DLT) of trabec | tedin give | en in association | with metron | onne |
| | and the dose cyclophospha | | (DLT) of trabec | tedin give | en in association | with metion | |
| | cyclophospha | | (DLT) of trabec | tedin give | en in association | with metron | |
| | cyclophospha<br>Definitions | amide. | | | | | |
| Enducinta | cyclophospha Definitions Dose-lim | amide. niting toxicity (DLT): | | | | | |
| Endpoints | cyclophospha Definitions Dose-lim | amide. niting toxicity (DLT): Il the criteria below: | : A DLT is defi | ned as an | AE or laboratory | | |
| Endpoints | cyclophospha Definitions Dose-lim fulfills al | niting toxicity (DLT): If the criteria below: Occurs during the | : A DLT is defi | ned as an | AE or laboratory reatment. | abnormality | |
| Endpoints | cyclophospha Definitions Dose-lim fulfills al | niting toxicity (DLT): If the criteria below: Occurs during the Is considered to learn | : A DLT is defi<br>e first cycle (4 w<br>be at least possib | ned as an<br>veeks) of to | AE or laboratory reatment. to the study treatm | abnormality | that |
| Endpoints | cyclophospha Definitions Dose-lim fulfills al | niting toxicity (DLT): Il the criteria below: Occurs during the Is considered to lead to the control of the | : A DLT is defi<br>e first cycle (4 w<br>be at least possib | ned as an<br>veeks) of to | AE or laboratory reatment. | abnormality | that |
| Endpoints | cyclophospha Definitions Dose-lim fulfills al | niting toxicity (DLT): If the criteria below: Occurs during th Is considered to l Meets one of th CTCAEv4.0: | : A DLT is defi<br>e first cycle (4 w<br>be at least possib<br>ne criteria below | ned as an<br>veeks) of to<br>oly related<br>w, graded | AE or laboratory reatment. to the study treatment as outlined or a | abnormality nent. | that<br>NCI |
| Endpoints | cyclophospha Definitions Dose-lim fulfills al | niting toxicity (DLT): If the criteria below: Occurs during the Is considered to lead to le | : A DLT is defi<br>e first cycle (4 w<br>be at least possib<br>ne criteria below<br>rade 4 toxicity | ned as an veeks) of to oly related w, graded | AE or laboratory reatment. to the study treatment as outlined or a for vomiting v | abnormality nent. | that<br>NCI |
| Endpoints | cyclophospha Definitions Dose-lim fulfills al | niting toxicity (DLT): If the criteria below: Occurs during the Is considered to lead to le | : A DLT is defi<br>e first cycle (4 w<br>be at least possib<br>ne criteria below | ned as an veeks) of to oly related w, graded | AE or laboratory reatment. to the study treatment as outlined or a for vomiting v | abnormality nent. | that<br>NCI |

1rst episode of nausea without maximal symptomatic/ prophylactic treatment and if toxicity is transaminitis, which may last > 7 days if total bilirubin is normal or grade =<1)

- Grade >= 3 hematologic toxicity lasting for > 7days
- Grade 4 neutropenia with fever
- Grade > 2 thrombocytopenia with bleeding
- Is unrelated to disease, disease progression, inter-current illness, or concomitant medications.

In addition, any AE related to treatment and considered as clinically significant on the opinion on the sponsor and of the investigators

- Maximum tolerated dose (MTD): the MTD is defined as the highest dose at which no more than 1 in 6 of the patients in the cohort experienced a DLT in the first treatment cycle.
- Recommended phase II dose (RP2D): will be identified by the steering committee based on the MTD, additional safety data (all cycles), PK and PD data. Data from all cycles will be used to define the dose level to be recommended for further investigations in phase II. An IDMC will be requested to assess safety data and validate the RP2D.

# Primary Endpoints:

- Toxicity graded using the common toxicity criteria from the NCI v4.0.
- Incidence rate of DLT at each dose level on cycle 1.

#### Secondary Endpoints:

- Objective response under treatment defined as complete (CR) or partial response (PR) as per RECIST v1.1 criteria. Objective response (CR or PR) under treatment is recorded from study treatment initiation until the end of treatment, with confirmation of responses ≥ 4 weeks after initial documentation, as per RECIST 1.1. Objective response under treatment is determined once all the data for the patient is known.
- 6-month non-progression defined as CR, PR or stable disease more than 24 weeks according to RECIST v1.1 criteria.
- 1-year Overall Survival (OS) defined as the time from study treatment initiation to death (of any cause).
- 1-year Progression-Free Survival (PFS) defined as the time from study treatment initiation to disease progression (defined as per RECIST v1.1) or death (of any cause), whichever occurs first.
- PK measurements expressed as the AUC, the half-life of trabectedin, CP and concentration peak.
- Pharmacodynamic study:
  - Blood: Serum/plasma cytokines levels (INFγ, TNFα, IL2,4,6,10) by ELISA; Serum/plasma VEGF and TPS-1 levels by ELISA, monocytes, Treg, CD4+, CD8+ and DR lymphocytes subpopulations monitoring, CD4+/CD8+ ratio (Flow Cytometry),
  - Tumor: Fresh pre-treatment and on-treatment tumor biopsies will be collected to assess pharmacodynamics changes of TAM infiltration and additional tumor markers. Frozen biopsy samples will be analyzed for:
    - Hematoxylin and eosin staining (H&E).
    - Immunohistochemistry (IHC) assessments include, but are not limited to the following markers: CSF-1R, CD68/CD163, CD68/MHC class II, CD31 (microvessel density), Ki67 and other exploratory markers. The analysis will be prioritized based on the amount of material available.

# Phase II trial:

#### Primary Endpoints:

- 6-month non-progression as defined above for the phase I escalation study.
- Disease status at 6 months will be reviewed by an expert radiologist. Reviewed data will be used for this primary endpoint analysis.

# Secondary Endpoints:

Toxicity, objective response under treatment, 1-year OS and 1-year PFS defined above for the phase I escalation study except for the PD study which is optional in this phase II trial.

#### **Sample Size Considerations:**

<u>Phase I (Dose escalation part):</u> based on a 3 + 3 traditional design with 4 dose levels with a minimum of 3 patients and a maximum of 6 patients per dose level: 24 eligible and assessable patients maximum will be needed.

Patients fulfilling the inclusion criteria will be enrolled in successive cohorts of 3 to 6 patients. If no DLT is observed during the first 4 weeks of study treatment in 3 patients, the dose of trabectedin will be escalated to the dose level (DL) immediately above. If One DLT is observed among 3 patients, the cohort will be expanded to 6 evaluable patients. If two patients out of 3 or 2 /6 patients experience a DLT, the dose will be considered intolerable and the DL immediately below will be further explored. The recommended phase II dose (RP2D) will be defined based on safety, PK data and PD data (optimal biological dose).

#### Phase II:

The EORTC suggest that 3 and 6-month non-progression rates (NPR) are relevant endpoints in STS phase II trials. We rely on an optimal two-stage Simon's design. Using unacceptable and acceptable 6-month non-progression rates of 20% and 40% respectively, a 5% type I error rate (bilateral), and a 20% type II error rate (80% power), a total of 43 eligible and assessable subjects will be necessary, with 13 subjects recruited to the first stage. At the end of the first stage, the trial will be terminated if 3 or less responses are observed. Otherwise, the second group of 30 subjects will be recruited, and a total of 13 responses or more will be required to claim activity of the drug. Assuming, 10% are not eligible or cannot be assessed for the primary endpoint, 47 patients will be recruited.

# **Definition of study populations**

#### Phase I trial

Population assessable for safety (primary analysis): all patients who completed the DLT assessment period or who developed DLT are included in the analysis.

# Patient's replacement

- If a patient cannot complete the full DLT evaluation period (28 days) and goes off-treatment for reasons other than toxicity, this patient can be replaced.
- Patients with DLT will never be replaced.
- All patients will be fully described in the analysis.
- Only patients who completed the DLT assessment period or who develop DLT are included in the analysis for escalation.

# Phase II trial

- Eligible population: All patients included without major violation of eligibility criteria.
- Population evaluable for efficacy:
  - All patients eligible and for whom the following conditions are satisfied:
    - O Diagnosis of STS at inclusion is confirmed after central review, except in case of diagnosis was reviewed in the RRePS Network,
    - For STS: Diagnosis of progressive disease at inclusion is confirmed after central review of the inclusion scans or MRI,
    - Received at least one administration of the treatment,
    - At least one disease measurement recorded not less than eight weeks after treatment onset.
- The following patients will also be included in the population evaluable for efficacy; they will be considered as failures for the primary endpoint (i.e. disease progression at six months for STS) and not be replaced in the primary efficacy analysis:
  - Any eligible patients who received at least one administration of the treatment and experienced disease progression or died due to disease progression prior to response evaluation (will be considered as an "early progression").
  - Patients withdrawn due to drug-related toxicity without any tumor assessments after the start of study treatment.
  - Patients who received at least one administration of the treatment AND withdrawn due to significant clinical deterioration of unknown reason AND without any tumor assessments after the start of study treatment.
- • Safety population: all patients having received at least one treatment administration.

#### Patient's replacement

# Statistical considerations

Any patient not eligible or not assessable for efficacy will be replaced.

However, any patient who received at least one administration of the study drug will be included in the safety analysis.

#### Statistical analysis

For the phase I trial, two documents will be produced by the statistician:

- A statistical analyse plan (SAP) before the first patient's inclusion,
- A statistical report.

For the phase II trial, four documents will be produced by the statistician:

- Two statistical analyse plans (SAP): one for the interim statistical analysis and one for the final statistical analysis.
- Two statistical reports: one for the interim statistical analysis and one for the final statistical analysis.

At the end of the phase I trial, an IDMC will be requested to assess safety data based on the statistical report produced by the statistician of the study. Similarly, an IDMC will be requested at the end of the first stage of the phase II trial to analyse preliminary safety and efficacy data.

# Patient characteristics at baseline

The patients entered into the study will be described according to the following characteristics:

- Compliance with eligibility criteria,
- Epidemiological characteristics,
- Clinical and laboratory characteristics,
- Treatment characteristics.

#### Endpoint analysis PHASE I trial

- Primary endpoint will be analyzed on the population assessable for safety of the phase I trial.
- Toxicity will be graded using the common toxicity criteria from the NCI v4.0.
- Incidence rate of DLT will be reported at each dose level on cycle 1.
- All analyses for the phase I trial will be descriptive; no p-values will be calculated. Data
  analyses will be provided by dose groups and for all study patients, combined wherever
  appropriate. For continuous variables, summary statistics will include number of patients,
  mean, median, standard deviation, standard error, minimum, and maximum. Categorical
  endpoints will be summarized using number of patients, frequency, percentages, and
  standard errors. Missing data will not be imputed.

# Endpoint analysis PHASE II trials

- Efficacy endpoints will be analyzed on the population assessable for efficacy.
- The safety analysis will be performed on the safety population.
- Quantitative variables will be described using mean and standard deviations if the normality assumption is satisfied, else other descriptive statistics (median, range, quartiles) will be reported.
- Qualitative variables will be described using frequency, percentage and 95% confidence interval (binomial law).
- Objective response rate under treatement, 6-month non-progression rate will be calculated using binomial estimates and reported with their 95% confidence interval (CI).
- Survival endpoints will be analysed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method. Multivariate analyses can also be carried out based on Cox's proportional risk method and after checking the risk proportionality hypothesis.

# Interim statistical analysis (phase II ONLY)

An interim statistical analysis will be carried out after the inclusion of the first 13 eligible and assessable patients. The trial will be terminated if 3 or less responses are observed. Otherwise, the second group of 30 subjects will be recruited. At the end of this first stage, an Independent Data Monitoring Committee (IDMC) will be request to analyze preliminary efficacy and safety data based on the statistical report produced by the statistician of the study. Inclusion will not be suspended during this interim analysis.

| | | | | S | chedule | of assess | sments a | nd proc | edures - | - Phase | I | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | CYC | | | | CYC | LE 2 | | | | CLE 3 | | CYCLE N | END OF TREATMEN |
| | SCREENING | Wk1 | Wk 2 | Wk3 | Wk 4 | Wk 5 | Wk 6 | Wk7 | Wk 8 | Wk9 | Wk 10 | Wk11 | Wk 12 | D1 to D7 | |
| CP b.i.d | | X | | X | | X | | X | | X | | X | | D15 to D21 | |
| Trabectedin i.v | | D1 | D8 | D15 | | D1 | D8 | D15 | | D1 | D8 | D15 | | D1, D8 and<br>D15 | |
| 24h-36h Hosp | | D1 | | D15 | | | | | | | | | | | |
| Ambulatory Hosp | | | D8 | | | D1 | D8 | D15 | | D1 | D8 | D15 | | D1, D8 and<br>D15 | |
| Consultation | X | | | | | | | | | | | | | | X |
| Informed consent | X | | | | | | | | | | A A | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | |
| Concomitant treatments | X | X | | | | | | | | X | | | | | |
| Physical exam | X | X | | X | | X | | | | X | | | | D1 | X |
| Vital signs | X | X | | X | | X | | | | X | | | | D1 | X |
| Height | X | | | | | | | A | | | | | | | |
| Weight | X | X | | X | | X | | | | X | | | | D1 | X |
| Performance status | X | X | | X | | X | | | | X | | | | D1 | X |
| Hematology <sup>a</sup> | X | X | X | X | | X | X | X | | X | X | X | | X <sup>d</sup> | X |
| Biochemistry <sup>b</sup> | X | X | X | X | · 1 | X | X | X | | X | X | X | | $X^{d}$ | X |
| ECG | X | X | | | | | | | | | | | | | X |
| Toxicity | | X | | | 4 | | | | | X | | | | | |
| Tumor measurement | X | | Repeated | every 8 we | eeks. Docu | mentation | (radiologic | e) must be | provided for | | removed from | m study for | progressive | disease | X |
| B-HCG <sup>c</sup> | X | X | | | | | | | | | | | | | |
| PK | | D1 | P. 4 | D15 | | | | | | | | | | | |
| Biomarkers | | X | | | | X | | | | | | | | | |
| Biopsy | | X | | | D28 | | | | | | | | | | |
| Echocardiography | X | | | | | | | | Repe | eated if ind | licated | | | | • |
| Serious and/ or non- serious<br>adverse events collection | X | | Repeated if indicated Throughout the study | | | | | | | | | | X (until 30 days later las<br>dose administered and<br>beyond this period only<br>SAEs related to research<br>or IMP) | | |

a: Hemoglobin, platelets, CBC w/diff

b: Albumin, Alkaline phosphatase, total bilirubin, bicarbonate, calcium, chloride, creatinine, CPK, glucose, LDH, phosphorus, potassium, total protein, SGOT [AST], SGPT [ALT], sodium

c: if indicated and repeated if necessary d: on weeks 1, 2 and 3 of each subsequent cycle

| | | | | So | chedule | of assess | ments a | nd proce | edures – | Phase I | I | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | CYC | | | | CYC | CLE 2 | | | | CLE 3 | | CYCLE N | END OF TREATMENT |
| | SCREENING | Wk1 | Wk 2 | Wk3 | Wk 4 | Wk 5 | Wk 6 | Wk7 | Wk 8 | Wk9 | Wk 10 | Wk11 | Wk 12 | D4 + D5 | |
| CP b.i.d | | X | | X | | X | | X | | X | | X | | D1 to D7<br>D15 to D21 | |
| Trabectedin i.v | | D1 | D8 | D15 | | D1 | D8 | D15 | | D1 | D8 | D15 | | D1, D8 and<br>D15 | |
| Ambulatory Hosp | | D1 | D8 | D15 | | D1 | D8 | D15 | | D1 | D8 | D15 | | D1, D8 and<br>D15 | |
| Consultation | X | | | | | | | | | | | | | 210 | X |
| Informed consent | X | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | 4 | | | | | | | |
| Concomitant treatments | X | X | | | | | | | | X | | | | | |
| Physical exam | X | X | | X | | X | | | | X | | | | D1 | X |
| Vital signs | X | X | | X | | X | | | | X | | | | D1 | X |
| Height | X | | | | | 4 | | | | | | | | | |
| Weight | X | X | | X | | X | | A | | X | | | | D1 | X |
| Performance status | X | X | | X | | X | P 4 | | | X | | | | D1 | X |
| Hematology <sup>a</sup> | X | X | X | X | | X | X | X | | X | X | X | | X <sup>d</sup> | X |
| Biochemistry <sup>b</sup> | X | X | X | X | | X | X | X | | X | X | X | | $X^d$ | X |
| ECG | X | | | | | | | | | | | | | | X |
| Toxicity | | X | | | | | | | | X | | | | | |
| Tumor measurement | X | | Repeated | every 8 w | eeks. Docu | mentation | (radiologic | e) must be | provided for | or patients | removed from | n study for | progressive | disease | X |
| B-HCG <sup>c</sup> | X | X | 4 | | | | | | | | | | | | |
| Biomarkers (optional) | | X | | | | X | | | | | | | | | |
| Biopsy (optional) | | X | P 4 | | D28 | | | | | | | | | | |
| Echocardiography | X | | | | | | | | Repe | eated if ind | icated | | | | |
| Serious and/ or non- serious adverse events collection | X | | | | | | | Througho | ut the stud | ly | | | | | X (until 30 days later last<br>dose administered and<br>beyond this period only<br>SAEs related to research<br>or IMP) |

a: Hemoglobin, platelets, CBC w/diff

PROT\_TARMIC\_V6.0|11|12|2018| Page 10 sur 11

b: Albumin, Alkaline phosphatase, total bilirubin, bicarbonate, calcium, chloride, creatinine, CPK, glucose, LDH, phosphorus, potassium, total protein, SGOT [AST], SGPT [ALT], sodium c: if indicated and repeated if necessary

d: on weeks 1, 2 and 3 of each subsequent cycle

